CLINICAL TRIAL: NCT03661021
Title: Study of the Ability of a New Technique to Effectively Diagnose Movement Disorders
Acronym: Sante-Fe
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Xin Xin Yu, MD, Physician, The Cleveland Clinic
Other Study IDs: Sante-Fe
Record Dates: First submitted 2018-08-09; First posted 2018-09-07 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-08

CONDITIONS: Functional Movement Disorder
Keywords: Functional movement disorder; Functional neurological disorder; FMD; Psychogenic movement disorder; Movement Disorders
MeSH Terms: conditions — Conversion Disorder; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Sante Fe is an investigation of a new technique to distinguish between different types of movement disorders, specifically organic versus functional, by observing changes in involuntary movements in two different situations.

DETAILED DESCRIPTION:
This study involves a short, one-time visit. Subjects will be asked to undergo a brief neurological examination while being video taped in two different scenarios. The severity of the abnormal movement will be analyzed and compared among subjects with functional (FMD) versus organic movement disorders (OrgMD).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a clinical diagnosis of Functional Movement Disorder (e.g. functional tremor, functional dystonia, functional myoclonus) based on Fahn-Williams criteria or OrgMD (e.g. Parkinson disease, essential tremor, cervical dystonia) evaluated by a fellowship-trained movement disorder neurologist at Cleveland Clinic
2. Patients with mild to severe involuntary movement as a result of the movement disorder, visible for video-recording.

Exclusion Criteria:

1. Significant cognitive impairment that prevents proper informed consent
2. Patients whose movement disorders cannot be captured on video

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Functional or Organic movement disorders at Cleveland Clinic Center for Neurological Restoration
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Change in Simplified Functional Movement Disorders Rating Scale (sFMDRS) score according to video raters between two conditions in FMD vs OrgMD patients. | Because this is a one-time visit study, outcome will be measured during the visit, data reported at study conclusion after successfully recruiting 40 subjects and completing analysis with projected finish date in 1 year
  Change in Simplified Functional Movement Disorders Rating Scale (sFMDRS) score according to video raters between two conditions in FMD vs OrgMD patients. Score reports total abnormal movement score ranging from 0-3 for 9 different regions of the body or body functions. Higher score implies more severe movement.

SECONDARY OUTCOMES:
The difference in the numerical change in self-perception of movement severity between two conditions in FMD vs OrgMD patients | Because this is a one-time visit study, outcome will be measured during the visit, data reported at study conclusion after successfully recruiting 40 subjects and completing analysis with projected finish date in 1 year
  The difference in the numerical change in self-perception of movement severity, as measured by a Likert-style scale, between two conditions in FMD vs OrgMD patients. Self-perception is scored on a scale of 0-4, with a higher score indicating more severe abnormal movement.

OTHER OUTCOMES:
Correlation between severity of depression or anxiety using PHQ-SADS scale and degree of change in severity of abnormal movement | Because this is a one-time visit study, outcome will be measured during the visit, data reported at study conclusion after successfully recruiting 40 subjects and completing analysis with projected finish date in 1 year
  Correlation between severity of depression or anxiety using PHQ-SADS scale and degree of change in severity of abnormal movement. Scale includes three sets of questions relating to symptoms of anxiety and depression. Each symptom is scored on a range of 0-2 or 3 and summed. Higher score indicates higher levels of anxiety or depression symptoms.
Correlation between health care utilization using Health Care Utilization scale and degree of change in severity of abnormal movement | Because this is a one-time visit study, outcome will be measured during the visit, data reported at study conclusion after successfully recruiting 40 subjects and completing analysis with projected finish date in 1 year
  Correlation between health care utilization using Health Care Utilization scale and degree of change in severity of abnormal movement. Scale asks about number of health care related experiences in the past 6 months.
Correlation between illness belief/diagnosis agreement using B-IPQ and Agreement with Diagnosis scales and degree of change in severity of abnormal movement | Because this is a one-time visit study, outcome will be measured during the visit, data reported at study conclusion after successfully recruiting 40 subjects and completing analysis with projected finish date in 1 year
  Correlation between illness belief/diagnosis agreement using B-IPQ and Agreement with Diagnosis scales and degree of change in severity of abnormal movement. B-IPQ asks subjects to answer questions about the impact of their illness on their lives on a scale of 0-10, where higher implies greater impact. Agreement with Diagnosis scale asks FMD subjects to rate the confidence in their diagnosis on a scale of 0-10, with 10 implying full confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Xin Yu, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hinson VK, Haren WB. Psychogenic movement disorders. Lancet Neurol. 2006 Aug;5(8):695-700. doi: 10.1016/S1474-4422(06)70523-3. PMID 16857575
- [Background] Voon V, Brezing C, Gallea C, Ameli R, Roelofs K, LaFrance WC Jr, Hallett M. Emotional stimuli and motor conversion disorder. Brain. 2010 May;133(Pt 5):1526-36. doi: 10.1093/brain/awq054. Epub 2010 Apr 5. PMID 20371508
- [Background] van Poppelen D, Saifee TA, Schwingenschuh P, Katschnig P, Bhatia KP, Tijssen MA, Edwards MJ. Attention to self in psychogenic tremor. Mov Disord. 2011 Dec;26(14):2575-6. doi: 10.1002/mds.23911. Epub 2011 Oct 24. No abstract available. PMID 22025317
- [Background] de Lange FP, Roelofs K, Toni I. Increased self-monitoring during imagined movements in conversion paralysis. Neuropsychologia. 2007 May 15;45(9):2051-8. doi: 10.1016/j.neuropsychologia.2007.02.002. Epub 2007 Feb 11. PMID 17367826
- [Background] Sitek EJ, Slawek J, Wieczorek D. [Self-awareness of deficits in Huntington's and Parkinson's disease]. Psychiatr Pol. 2008 May-Jun;42(3):393-403. Polish. PMID 19899567
- [Background] Amanzio M, Monteverdi S, Giordano A, Soliveri P, Filippi P, Geminiani G. Impaired awareness of movement disorders in Parkinson's disease. Brain Cogn. 2010 Apr;72(3):337-46. doi: 10.1016/j.bandc.2009.10.011. Epub 2009 Nov 14. PMID 19914762
- [Background] Straumann C, Anderson JR. Mirror-induced social facilitation in stumptailed macaques (Macaca arctoides). Am J Primatol. 1991;25(2):125-132. doi: 10.1002/ajp.1350250206. PMID 31948184
- [Background] Landers DM, McCullagh PD. Social facilitation of motor performance. Exerc Sport Sci Rev. 1976;4:125-62. No abstract available. PMID 798687
- [Background] Nielsen G, Ricciardi L, Meppelink AM, Holt K, Teodoro T, Edwards M. A Simplified Version of the Psychogenic Movement Disorders Rating Scale: The Simplified Functional Movement Disorders Rating Scale (S-FMDRS). Mov Disord Clin Pract. 2017 Mar 11;4(5):710-716. doi: 10.1002/mdc3.12475. eCollection 2017 Sep-Oct. PMID 30363505